CLINICAL TRIAL: NCT00331071
Title: Postmarketing Study of ORTHO EVRA in Relation to Venous Thromboembolism, Ischemic Stroke, and Myocardial Infarction
Brief Title: Postmarketing Study of ORTHO EVRA (Norelgestromin and Ethinyl Estradiol Contraceptive Patch) in Relation to Venous Thromboembolism (Blood Clots), Stroke and Heart Attacks
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Boston Collaborative Drug Surveillance Program (Other)
Responsible Party: Sponsor
Other Study IDs: CR012025; BCDSP-01
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Contraception; Female Contraception
Keywords: Contraception; Hormonal contraception; Oral contraception; Ethinyl estradiol, Progestin, Contraception; Transdermal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 001: Ortho Evra transdermal patch containing 6 mg NGMN/0.75 mg EE worn for 1 week and replaced for 3 consecutive weeks fourth week is patch free
  Interventions: Drug: Ortho Evra transdermal patch containing 6 mg NGMN/0.75 mg EE
- 002: Monophasic or triphasic Oral contraceptive tablet 35 mcg EE for 21 consecutive days followed by no or drug-free tablet for 7 days
  Interventions: Drug: Monophasic or triphasic Oral contraceptive tablet

INTERVENTIONS:
Drug: Monophasic or triphasic Oral contraceptive tablet — fourth week is patch free
  Groups: 002
Drug: Ortho Evra transdermal patch containing 6 mg NGMN/0.75 mg EE — worn for 1 week and replaced for 3 consecutive weeks
  Groups: 001

SUMMARY:
The purpose of the study is to assess the occurrence of venous thromboembolism (blood clots), stroke, and heart attack in current users of ORTHO EVRA compared to current users of norgestimate-containing oral contraceptives with 35 mcg ethinyl estradiol with special attention to duration of use. The study uses data from the PharMetrics Patient-Centric Database and MarketScan database, which are US medical claims databases.

DETAILED DESCRIPTION:
ORTHO EVRA is a newly developed transdermal (absorbed through the skin) contraceptive (birth control) system (a "patch") available in the U.S. since April 2002. The study uses data from the PHARMetrics and MarketScan databases to assess the occurrence of venous thromboembolism (blood clots), ischemic stroke (blockage of an artery that supplies blood to the brain), and acute myocardial infarction (heart attack) in current first time users of ORTHO EVRA compared to current first time users of norgestimate-containing oral (by mouth) contraceptives with 35 mcg ethinyl estradiol. The PHARMetrics database is an ongoing longitudinal database with information on about 17 million people. It is made up of data contributed by managed care plans in the United States and contains information on paid claims for pharmaceuticals, medical diagnoses and procedures, and demographic (age, race, etc) information. There will be 3 sets of cases reflecting women who have a first-time recorded claim for an ICD-9 (International Classification of Diseases , ninth revision) diagnosis during the study period (a) venous thrombosis or pulmonary embolism (blood clot in the lung) with hospitalization during the study period and who had subsequent claims for anticoagulant treatment, (b) ischemic stroke and who were hospitalized, (c) acute myocardial infarction or acute coronary revascularization (restoration of blood supply to the heart) and who were hospitalized. Three separate sets of controls (patients) will be identified for each outcome. One analysis will estimate the relative risk of idiopathic (of unknown cause) ischemic stroke or myocardial infarction, and another analysis will estimate the relative risk of idiopathic venous thromboembolism (deep vein thrombosis or pulmonary embolism). A specific analysis called a "Conditional logistic regression" (conditional on the matching factors) will be used in this study. Analyses will be stratified by calendar year. The analyses will be repeated including non-idiopathic (ie, of known cause) cases of venous thromboembolism, stroke, and heart attacks. The original study runs through March 2005, with updates to through August 2006, and October 2007. A transdermal patch containing 6 mg norelgestromin (NGM) and 0.75 mg ethinyl estradiol (EE) is worn for 1 week and replaced weekly for 3 consecutive weeks; the fourth week is patch-free. Monophasic (all pills have the same hormones at the same concentration) or triphasic (3 different pills are taken during the cycle) oral contraceptive pill is taken for 21 consecutive days followed by no pill or a drug-free pill for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Users of Ortho Evra or first time users of norgestimate-containing oral contraceptives with 35 mcg ethinyl estradiol between April 1, 2002 and December 31, 2004, who are identified in the PHARMetrics database using the National Drug Code (NDC) assigned by the FDA and modified by Pharmetrics
* 6 months of enrollment in a health plan prior to the event date of their matched case
* Start of study contraceptive use after January 1, 2002
* Updates to the original study included users of Ortho Evra or first time users of norgestimate-containing oral contraceptives identified in the PHARMetrics database and a US healthcare claims database through August 2006 and October 2007

Exclusion Criteria:

* Patients with any ICD-9 code for cancer (except for non-melanoma skin cancer), renal failure, or chronic inflammatory disease

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Data collected from PharMetrics, a United States based, ongoing longitudinal database of data contributed by managed care plans that contains information on unpaid claims for pharmaceuticals, medical diagnoses and procedures and from MarketScan database, a US health care claims database.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2002-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
First-time recorded claim for a) venous thrombosis or pulmonary embolism with hospitalization and claims for anticoagulant treatment, b) ischemic stroke/hospitalized, c) acute myocardial infarction or acute coronary revascularization/hospitalized | Throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Jick SS, Kaye JA, Russmann S, Jick H. Risk of nonfatal venous thromboembolism in women using a contraceptive transdermal patch and oral contraceptives containing norgestimate and 35 microg of ethinyl estradiol. Contraception. 2006 Mar;73(3):223-8. doi: 10.1016/j.contraception.2006.01.001. Epub 2006 Jan 26. PMID 16472560
- See also: Postmarketing Study of ORTHO EVRA in Relation to Non-Fatal Venous Thromboembolism and Cerebral Sinus Thrombosis-September 21, 2005 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=739&filename=CR012025_CSRa.pdf
- See also: Postmarketing Study of ORTHO EVRA in Relation to Ischemic Stroke, Acute Myocardial Infarction and Cerebral Sinus Thrombosis-December 15, 2005 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=739&filename=CR012025_CSRb.pdf
- See also: Postmarketing Study of ORTHO EVRA in Relation to Non-Fatal Venous Thromboembolism-January 16, 2007 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=739&filename=CR012025_CSRc.pdf
- See also: Report on the 2007 Update on Post marketing Study of ORTHO EVRA in Relation to Non-Fatal Venous Thromboembolism, Ischemic Stroke, Acute Myocardial Infarction, and Cerebral Vascular Sinus Thrombosis-May 20, 2008 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=739&filename=CR012025_CSRd.pdf